CLINICAL TRIAL: NCT00524446
Title: A Single-centre, Randomised, Single-blind, Parallel Group Clinical Trial in Rural Malawi, Testing the Growth Promoting Effect of Long-term Complementary Feeding of Infants With a High-energy, Micronutrient Fortified Spread
Brief Title: Controlled Trial to Test the Efficacy of Lipid-based Nutrient Supplements to Prevent Severe Stunting Among Infants
Acronym: LCNI-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Academy of Finland (Other); Foundation for Paediatric Research, Finland (Other); Medical Research Fund of the Tampere University Hospital, Finland (Other)
Responsible Party: Principal Investigator, Per Ashorn, Professor of International Health, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTS-2007-02-19
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Malnutrition; Stunting; Developmental Delay
Keywords: Infant; Sub-Saharan Africa; Complementary feeding; Fortified spread; Lipid-based nutrient supplement; Malnutrition; Stunting; Growth; Morbidity; Development; Haemoglobin
MeSH Terms: conditions — Malnutrition; Growth Disorders; Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ST-DI (No Intervention): Standard treatment - delayed intervention. Counselling on complementary feeding + Vitamin A (200,000 IU) every 6 months until 36 months + 1 kg maize / soy flour 2-weekly (71 g / day) between 18 and 30 months of age.
- FSm (Experimental): Fortified Spread (milk). Counseling + Vitamin A as for ST-DI + 750 g of fortified spread (FSm) 2-weekly (54 g / day) between 6 and 18 months of age.
  Interventions: Dietary Supplement: Milk-containing fortified spread
- FSs (Experimental): Counselling + Vitamin A as for ST-DI + 750 g of modified fortified spread (FSs) 2-weekly (54 g / day) between 6 and 18 months of age.
  Interventions: Dietary Supplement: Soy-containing fortified spread
- LP (Experimental): Likuni Phala. Counseling + Vitamin A as for ST-DI + 1 kg fortified maize / soy flour 2-weekly (71 g / day) between 6 and 18 months of age.
  Interventions: Dietary Supplement: Maize-soy flour

INTERVENTIONS:
Dietary Supplement: Milk-containing fortified spread — Counseling + Vitamin A as for ST-DI + 750 g of fortified spread (FSm) 2-weekly (54 g / day) between 6 and 18 months of age.
  Arms: FSm
Dietary Supplement: Soy-containing fortified spread — Counseling + Vitamin A as for ST-DI + 750 g of modified fortified spread (FSs) 2-weekly (54 g / day) between 6 and 18 months of age.
  Arms: FSs
Dietary Supplement: Maize-soy flour — Counseling + Vitamin A as for ST_DI + 1 kg fortified maize / soy flour 2-weekly (71 g / day) between 6 and 18 months of age.
  Arms: LP

SUMMARY:
This study tests the hypothesis that infants receiving milk-powder containing fortified spread (lipid-based nutrient supplement) as a complementary food for one year have lower incidence of severe stunting (poor length gain) than infants who are provided with no extra food supplements or maize-soy flour for complementary porridge.

DETAILED DESCRIPTION:
Poor growth and severe childhood stunting is very common in rural Malawi and elsewhere in Sub-Sahara Africa. To date, few interventions have proven successful in promoting linear growth in early childhood. Our preliminary results from Malawi suggest that a year-long daily complementary feeding of infants with a high-energy, micronutrient-fortified spread (FS) may markedly reduce the incidence of severe stunting before the age of 18 months. In the present study the investigators will more carefully analyze the efficacy in linear growth promotion and other health benefits of this product when provided as a complementary food to infants between 6 and 18 months of age.

The study will be conducted in Lungwena area, Mangochi District, rural Malawi. Six-month old healthy infants are identified through community surveys in the study area. 840 infants meeting set criteria are randomized into receiving the following intervention between 6 and 18 months of age: 1) standard treatment ie no extra food supplements (but dietary supplementation between 18 and 30 months of age) (ST-DI, control group), 2), "standard" fortified spread with milk-powder as the protein source (FSm), 3) modified fortified spread with soy-powder as the protein source (FSs), or 4) fortified maize-soy flour (likuni phala, LP). The families receive the food supplements at 2-weekly intervals and the participants undergo an anthropometric and developmental evaluation and laboratory analyses at 12-week intervals. Outcome analyses are done at 18 and at 36 months of age.

The impact of the dietary interventions will be primarily assessed by comparing the incidence of severe stunting in the four study groups. Secondary outcomes include a number of anthropometric variables, morbidity, developmental milestones, and laboratory parameters. The study will also produce descriptive data on possible mechanisms for growth failure among the trial subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one guardian
* Age 5.50 months to 6.49 months
* Availability during the period of the study.
* Permanent resident of Lungwena Health Centre or Malindi Hospital catchment area

Exclusion Criteria:

* Existing or imminent severe stunting (HAZ < -2.8)
* Weight for length (WFH) < 80% of the reference median or presence of oedema
* Severe illness warranting hospital referral.
* History of allergy towards peanut
* History of anaphylaxis or serious allergic reaction to any substance, requiring emergency medical care
* Concurrent participation in any other clinical trial

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Incidence of severe stunting (Length-for-age Z score < -3) | 1 year after enrolment
Incidence of serious and non-serious adverse events | 1 year

SECONDARY OUTCOMES:
Incidence of moderate or severe stunting (Length-for-age Z-score < -2) | 1 year
Length gain (cm) | 1 year
Weight gain (g) | 1 year
Change in anthropometric indices (Weight-for-age Z-score, Weight-for-length Z-score, Length-for-age Z-score), mid-upper arm circumference and head circumference | 1 year
Incidence of moderate or severe underweight or wasting (Weight-for-age Z-score or Weight-for-length Z-score <-2 / -3 SD units) | 1 year
Blood haemoglobin, serum ferritin, vitamin A, and zinc concentration | 18 months of age
Motor, social, and language development (timing of acquisition of defined skills) | 1 year
Incidence of febrile illnesses and laboratory diagnosed malaria | 1 year
Morbidity for respiratory infections, diarrhea, and other illnesses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Study Director — University of Tampere Medical School, Finland; Kenneth Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- College of Medicine, University of Malawi, Mangochi, Malawi

REFERENCES:
- [Derived] Xu G, Davis JC, Goonatilleke E, Smilowitz JT, German JB, Lebrilla CB. Absolute Quantitation of Human Milk Oligosaccharides Reveals Phenotypic Variations during Lactation. J Nutr. 2017 Jan;147(1):117-124. doi: 10.3945/jn.116.238279. Epub 2016 Oct 19. PMID 27798342
- [Derived] Aakko J, Grzeskowiak L, Asukas T, Paivansade E, Lehto KM, Fan YM, Mangani C, Maleta K, Ashorn P, Salminen S. Lipid-based Nutrient Supplements Do Not Affect Gut Bifidobacterium Microbiota in Malawian Infants: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):610-615. doi: 10.1097/MPG.0000000000001333. PMID 27403608
- [Derived] Mangani C, Ashorn P, Maleta K, Phuka J, Thakwalakwa C, Dewey K, Manary M, Puumalainen T, Cheung YB. Lipid-based nutrient supplements do not affect the risk of malaria or respiratory morbidity in 6- to 18-month-old Malawian children in a randomized controlled trial. J Nutr. 2014 Nov;144(11):1835-42. doi: 10.3945/jn.114.196139. Epub 2014 Sep 17. PMID 25332483
- [Derived] Grzeskowiak L, Collado MC, Mangani C, Maleta K, Laitinen K, Ashorn P, Isolauri E, Salminen S. Distinct gut microbiota in southeastern African and northern European infants. J Pediatr Gastroenterol Nutr. 2012 Jun;54(6):812-6. doi: 10.1097/MPG.0b013e318249039c. PMID 22228076
- See also: College of Medicine homepage — http://www.medcol.mw/